CLINICAL TRIAL: NCT04301622
Title: Post Market Clinical Follow-Up Study for EVOLUTION® BIOFOAM® Tibia and EVOLUTION® CS/CR Porous Femur With Cruciate Sacrificing Inserts
Brief Title: Post Market Clinical Follow-Up Study for EVOLUTION® BIOFOAM® Tibia and EVOLUTION® CS/CR Porous Femur
Status: Active, not recruiting | Type: Observational
Sponsor: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 17K001
Record Dates: First submitted 2020-03-05; First posted 2020-03-10 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Knee Osteoarthritis; Traumatic Arthritis of Knee; Avascular Necrosis; Degenerative Joint Disease of Knee; Rheumatoid Arthritis of Knee; Correction of Functional Deformity
MeSH Terms: conditions — Osteoarthritis, Knee; Osteonecrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Primary Knee implants — Primary knee arthroplasty

SUMMARY:
MicroPort (MPO) is conducting this PMCF study to evaluate the safety and effectiveness of its EVOLUTION® BIOFOAM® Tibia and EVOLUTION® Cruciate Sacrificing/Cruciate Retaining (CS/CR) Porous Femur components, including EVOLUTION® CS tibial inserts. This type of study is required by regulatory authorities for all devices that have been approved in Europe to evaluate the medium and long-term clinical evidence.

DETAILED DESCRIPTION:
The objectives of this study are:

1. To estimate the individual component survivorship of EVOLUTION® BIOFOAM® Tibia and EVOLUTION® CS/CR Porous Femur components, including EVOLUTION® CS tibial inserts
2. To find out the cumulative incidence of component revision of each component in this combination.
3. To find out the functional outcome scores at early, midterm, and long term follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Has previously undergone or currently has determined to undergo a primary TKA with the specified combination of components: EVOLUTION® CS/CR Porous Femur, EVOLUTION® CS Tibial Insert, and EVOLUTION® BIOFOAM® Tibia and modular keel
2. Has previously undergone or currently has determined to undergo a primary TKA for any of the following:

   * non-inflammatory degenerative joint disease including osteoarthritis, traumatic arthritis, or avascular necrosis;
   * inflammatory degenerative joint disease including rheumatoid arthritis;
   * correction of functional deformity;
   * willing and able to complete required study visits and assessments through the 10 year postoperative follow-up visit.
3. Previously implanted subjects must be enrolled within 3 years (+6 months) of their primary TKA implantation

Exclusion Criteria:

1. Skeletally immature (less than 21 years of age) at time of implantation
2. Has or had an overt infection at the time of implantation
3. Has or had a distant foci of infections (which may cause hematogenous spread to the implant site) at the time of implantation
4. Has or had a rapid disease progression as manifested by joint destruction or bone absorption apparent on roentgenogram at the time of implantation
5. Has or had inadequate neuromuscular status (e.g., prior paralysis, fusion, and/or inadequate abductor strength), poor bone stock, poor skin coverage around the joint which would make the procedure unjustifiable
6. Has had a revision procedure(s) where other treatments or devices have failed; and treatment of fractures that are unmanageable using other techniques
7. Currently enrolled in another clinical investigation which could affect the endpoints of this protocol
8. Unwilling or unable to sign the Informed Consent document
9. Has documented substance abuse issues
10. Has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study
11. Currently incarcerated or has impending incarceration
12. Has a medical condition, as judged by the Investigator, that would interfere with the subject's ability to comply with the requirements of the protocol

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary TKA or Single study group with newly or previously implanted patients with EVOLUTION® BIOFOAM® Tibia and EVOLUTION® CS/CR Porous Femur with Cruciate Sacrificing Insert
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2032-02 (Estimated); Study Completion 2032-08 (Estimated)

PRIMARY OUTCOMES:
Individual component survivorship | 10 years post-operative
  Individual component survivorship for tibial base, femoral, and tibial CS insert at specified intervals out to 10 years follow-up.

SECONDARY OUTCOMES:
Patient Reported Outcomes- Knee Injury and Osteoarthritis Outcome Scores | 10 years post-operative
  -functional scores for subjects, as assessed by Knee Injury and Osteoarthritis Outcome Score (KOOS), out to 10 years follow-up
Patient Reported Outcomes- EuroQol-5D-5L Scores | 10 years post-operative
  -functional scores for subjects, as assessed by EuroQol-5D-5L (EQ-5D-5L) Scores, out to 10 years follow-up
Patient Reported Outcomes- Forgotten Joint Score | 10 years post-operative
  -subject satisfaction measures with their Total Knee Arthroplasty (TKA) procedure using the Forgotten Joint Score
Patient Reported Outcomes- Satisfaction Survey | 10 years post-operative
  -subject satisfaction measures with their Total Knee Arthroplasty (TKA) procedure using the Satisfaction Survey
Incidence of component revision | 10 years post-operative
  the cumulative incidence of component revision at specified intervals will be determined out to 10 years follow-up
Radiolucencies | 10 years post-operative
  the presence, zone, and the size of radiolucencies surrounding implanted components will be determined
Adverse Events and Adverse Device Effects | 10 years post-operative
  characterization of adverse events and adverse device effects

CONTACTS AND LOCATIONS:
Overall Officials: Brian de Beaubien, MD, Principal Investigator — Covenant Medical Center
Locations (1):
- Covenant Medical Center, Saginaw, Michigan, United States

IPD SHARING:
Plan to Share IPD: No